CLINICAL TRIAL: NCT06514352
Title: The Effect of Skin-to-Skin Contact Based on Clinical Guidelines on Newborn Stress and Breastfeeding Success
Brief Title: The Effect of Skin-to-Skin Contact Based on Clinical Guidelines
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Principal Investigator, Tugce Sonmez, Principal Investigator, Gaziantep Islam Science and Technology University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 3304skincontact
Record Dates: First submitted 2024-07-09; First posted 2024-07-23 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2024-07

CONDITIONS: Breastfeeding; Newborn
Keywords: skin to contact; breastfeeding; newborn
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- skin-to-skin contact group immediately after birth (Experimental): The newborn is placed face to face on the mother's abdomen or chest in the first minute after birth. If medically necessary, suctioning can be done while on the mother's abdomen or chest and the baby is dried thoroughly. To prevent heat loss, the baby's back is covered with a pre-warmed blanket and a hat is placed on his head. All other interventions with the newborn can be postponed until at least the end of the first hour after birth or the first successful breastfeeding.
  Interventions: Other: Skin contact immediately after birth
- very early skin contact group (Experimental): In the first 30-40 minutes after birth, after the first and emergency intervention is given to the newborn in need of intervention, the newborn is placed face down on the mother's bare chest, naked with or without a hat. The newborn's back can be covered with a blanket.
  Interventions: Other: Very Early Skin contact
- early skin contact group (Experimental): It can start any time between the first hour and 24 hours after birth. The baby is naked (with or without a diaper) and placed face down on the mother's bare chest between the breasts. The mother can wear a blouse or shirt that opens at the front, or a hospital gown that can be tied at the back. The baby is placed inside the apron so that only the head is exposed. What the mother wears, how the baby is kept warm, and what is placed on the baby's back may vary. The most important thing is that the mother and baby are in direct skin-to-skin contact and the baby is kept dry and warm.
  Interventions: Other: Early Skin contact
- control group (No Intervention): No treatment will be performed on the mothers and newborns in the control group, and the hospital's routine practices (birthing support, newborn and maternal care) will be carried out.

INTERVENTIONS:
Other: Skin contact immediately after birth — In the immediate skin-to-skin contact group after birth, if the newborn does not need any intervention, he will be placed on the mother's chest immediately (without cord clamping) and skin-to-skin contact will begin. An average of 60 minutes of skin contact will be made until the first breastfeeding occurs. All routine practices for the newborn in the delivery room (except weight measurement) will be performed on the mother's chest. (n=48)
  Arms: skin-to-skin contact group immediately after birth
Other: Very Early Skin contact — In the very early skin-to-skin contact group, skin-to-skin contact will begin within the first 30-40 minutes after birth, after the first and emergency intervention is given to the newborn in need of intervention, and skin-to-skin contact will be carried out for an average of 60 minutes until the first breastfeeding occurs.(n=48)
  Arms: very early skin contact group
Other: Early Skin contact — For newborns who need intervention after birth and whose skin-to-skin contact cannot be started in the delivery room, skin-to-skin contact will begin within the first 24 hours after birth, after the newborn becomes stable.(n=48)
  Arms: early skin contact group

SUMMARY:
Newborn health indicators are important data that provide information about the welfare level of countries. Health professionals and relevant institutions have important responsibilities in protecting, developing and ensuring the continuity of newborn health. Health professionals use evidence-based practices revealed by scientific studies in their care approaches. Care and follow-up immediately after birth are very important. When the investigators look at the neonatal mortality rate in our country in 2019, it is shown as 5.3 per thousand and 5 per thousand in 2020. Therefore, neonatal-specific programs and practices need to be strengthened in order to reduce both neonatal and postneonatal death rates.

Midwives are the professional group that is with both the mother and the newborn during the birth and postpartum period, can initiate breastfeeding in the early period, and ensure optimal continuation of breastfeeding.

It is very important that the basic health indicators of the newborn improve and that the mother and newborn are monitored at certain standards during and after birth. These monitoring must be done according to the criteria. Genç et al. in 2022 to initiate and maintain skin-to-skin contact with the newborn during the postpartum period. (2023) skin-to-skin contact will be made between the mother and the newborn in accordance with the "Skin-to-Skin Contact and Kangaroo Care Clinical Practice Guide".

DETAILED DESCRIPTION:
Newborn health indicators are important data that provide information about the welfare level of countries. Health professionals and relevant institutions have important responsibilities in protecting, developing and ensuring the continuity of newborn health. Health professionals use evidence-based practices revealed by scientific studies in their care approaches. Care and follow-up immediately after birth are very important. When the investigators look at the neonatal mortality rate in our country in 2019, it is shown as 5.3 per thousand and 5 per thousand in 2020. Therefore, neonatal-specific programs and practices need to be strengthened in order to reduce both neonatal and postneonatal death rates.

Midwives are the professional group that is with both the mother and the newborn during the birth and postpartum period, can initiate breastfeeding in the early period, and ensure optimal continuation of breastfeeding.

It is very important that the basic health indicators of the newborn improve and that the mother and newborn are monitored at certain standards during and after birth. These monitoring must be done according to the criteria. Genç et al. in 2022 to initiate and maintain skin-to-skin contact with the newborn during the postpartum period. (2023) skin-to-skin contact will be made between the mother and the newborn in accordance with the "Skin-to-Skin Contact and Kangaroo Care Clinical Practice Guide".

Skin-to-skin contact (SC) is the placement of the baby on the mother's chest for at least one hour at birth or immediately after birth. A healthy, full-term baby who receives SC after birth directs himself to his mother's breast and nipple and starts sucking for about an hour. This application has many benefits for mother and baby. If the investigators look at the benefits for the mother; earlier separation of the placenta, reduced postpartum bleeding, increased breastfeeding self-efficacy, and reduced maternal stress levels. In addition, the increase in the mother's oxytocin level in the first hour after birth ensures the development and strengthening of bonding between mother and baby. The benefits for the baby are; These include reducing the negative consequences that may develop due to birth stress, effective thermoregulation, crying less and for a shorter period of time, reducing the likelihood of apnea, less physiological weight loss, and less stress response to painful procedures. At the same time, while SC reduces the rate of formula supplementation in the hospital, it has been shown to increase the initiation of breastfeeding and the level of exclusive breastfeeding, leading to a successful first breastfeeding and optimal breastfeeding.

SC application time and durations vary. SC at birth or immediately after birth: The newborn is placed face to face on the mother's abdomen or chest within the first minute after birth. If medically necessary, suctioning can be done while on the mother's abdomen or chest and the baby is dried thoroughly. To prevent heat loss, the baby's back is covered with a pre-warmed blanket and a hat is placed on his head. All other interventions with the newborn can be postponed until at least the end of the first hour after birth or the first successful breastfeeding.

Very early SC: Within the first 30-40 minutes after birth, after the first and emergency intervention is given to the newborn in need of intervention, the newborn is placed face down on the mother's bare chest, naked with or without a hat. The newborn's back can be covered with a blanket.

Early SC: It can begin any time between the first hour and 24 hours after birth. The baby is naked (with or without a diaper) and placed face down on the mother's bare chest between the breasts. The mother can wear a blouse or shirt that opens at the front, or a hospital gown that can be tied at the back. The baby is placed inside the apron so that only the head is exposed. What the mother wears, how the baby is kept warm, and what is placed on the baby's back may vary. The most important thing is that the mother and baby are in direct skin-to-skin contact and the baby is kept dry and warm.

A thesis study was planned to examine the relationship between skin-to-skin contact, which will be applied within the framework of these application timings, and neonatal stress and suckling success.

The thesis study was planned as a randomized controlled experimental study. The thesis is planned to be carried out at Tarsus State Hospital Maternity Room between August 2024 and January 2025.

The population of the study will be women who applied to Tarsus State Hospital Maternity Room for birth between the dates of the study. The sample consists of 48 (group 1 - sc immediately after birth), 48 (group 2 - very early sc), 48 (group 3 - early sc), 48 control group, who met the selection criteria, agreed to participate in the thesis study and were determined by power analysis. It will consist of a total of 192 women.

As data collection tools, socio-demographic characteristics introduction and questionnaire for skin contact and breastfeeding process, Skin Contact and Breastfeeding Process Follow-up Form, LATCH Breastfeeding Diagnosis Measurement Tool and Newborn Stress Scale will be used.

Socio-Demographic Characteristics Introduction and Questionnaire for Skin Contact and Breastfeeding Process: The form prepared by the researchers consists of 22 questions regarding the socio-demographic characteristics of the mothers and their spouses, the obstetric characteristics of the mothers and the newborn.

Skin Contact and Breastfeeding Process Follow-up Form: The form was created by researchers. This is the form in which information about the time when mothers start to apply skin-to-skin contact, the duration of skin-to-skin contact, the time to start breastfeeding, the duration of breastfeeding and the time for the baby to settle on the breast will be recorded.

LATCH Breastfeeding Diagnostic Measurement Tool: Breastfeeding status of mothers in the intervention and control groups in the postpartum period will be evaluated using the LATCH scale. LATCH Breastfeeding Diagnostic Measurement Tool was developed in 1986 by observing breastfeeding by healthcare professionals or researchers in the clinic; It is an assessment tool that is quick and easy to apply and was created to detect problems that may occur in breastfeeding. Scoring is between 0-2 and the maximum score that can be obtained is 10. In the measurement tool that does not have a cut-off point, a high score indicates that breastfeeding is successful. The reliability study was conducted by Adams and Hewell in 1997. The Turkish reliability study of the scale was conducted by Yenal and Okumuş (2003) and the Chronbach alpha value was found to be 0.95.

Newborn Stress Scale: The Newborn Stress Scale, developed by Ceylan and Bolışık (2017) to evaluate the stress level in premature babies, is suitable for use in term babies. Scale items were collected in 8 subgroups in a 3-point Likert type, including facial expression, body color, respiration, activity level, consolability, muscle tone, extremities, and posture. In scoring, each subgroup is evaluated between 0-2 points.

A minimum of 0 points and a maximum of 16 points are taken from the scale. As the score increases, the baby's stress level increases. Cronbach's alpha coefficient has been reported to be between 0.65-0.81.

Application Steps Group 1- SC Immediately After Birth: In the immediate skin-to-skin contact group after birth, if the newborn does not need any intervention, it will be placed on the mother's chest immediately (without cord clamping) and skin-to-skin contact will begin. An average of 60 minutes of skin contact will be made until the first breastfeeding occurs. All routine practices for the newborn in the delivery room (except weight measurement) will be performed on the mother's chest.

Group 2- Very Early SC: In the very early SC group, skin-to-skin contact will begin within the first 30-40 minutes after birth, after the first and emergency intervention is given to the newborn in need of intervention, and skin-to-skin contact will be carried out for an average of 60 minutes until the first breastfeeding occurs.

Group 3- Early SC: For the newborn who needs intervention after birth and for whom skin-to-skin contact cannot be started in the delivery room, skin-to-skin contact will begin within the first 24 hours after birth, after the newborn becomes stable.

Control group: No treatment will be performed on the mothers and newborns in the control group, and the hospital's routine practices will be carried out.

Newborn stress and LATCH score will be evaluated at the 12th and 24th hours after birth in all groups.

ELIGIBILITY:
Inclusion Criteria:

* Giving birth vaginally
* Primiparous pregnant
* Giving birth at 37 weeks or more
* Single and alive fetus
* Not being pregnant at risk
* Not being an individual with special needs
* Ability to communicate with the pregnant woman
* Stay in the neonatal intensive care unit for less than 24 hours

Exclusion Criteria:

* Having multiple pregnancies,
* Women who gave up participating in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Question Form for Socio-Demographic Characteristics Introduction and Skin Contact and Breastfeeding Process | immediately before intervention
  The form prepared by the researchers consists of 22 questions regarding the socio-demographic characteristics of the mothers and their spouses, the obstetric characteristics of the mothers and the newborn.
Skin Contact and Breastfeeding Process Follow-up Form | immediately after the intervention
  The form was created by researchers. This is the form in which information about the time when mothers start to apply skin-to-skin contact, the duration of skin-to-skin contact, the time to start breastfeeding, the duration of breastfeeding and the time for the baby to settle on the breast will be recorded.
LATCH Breastfeeding Diagnostic Measurement Tool | immediately after the intervention, 12 hours after birth, 24 hour after birth
  During the postpartum period, the breastfeeding status of mothers in the intervention and control groups will be evaluated using the LATCH scale. LATCH Breastfeeding Diagnostic Measurement Tool was developed in 1986 by observing breastfeeding by healthcare professionals or researchers in the clinic; It is an assessment tool that is quick and easy to apply and was created to detect problems that may occur in breastfeeding. Scoring is between 0-2 and the maximum score that can be obtained is 10. In the measurement tool that does not have a cut-off point, a high score indicates that breastfeeding is successful. The reliability study was conducted by Adams and Hewell in 1997. The Turkish reliability study of the scale was conducted by Yenal and Okumuş (2003) and the Chronbach alpha value was found to be 0.95.
Newborn Stress Scale | immediately after the intervention, 12 hours after birth, 24 hour after birth
  Newborn Stress Scale: The Newborn Stress Scale, developed by Ceylan and Bolışık (2017) to evaluate the stress level in premature babies, is suitable for use in term babies. The scale items were collected in 8 subgroups in a 3-point Likert type, including facial expression, body color, respiration, activity level, consolability, muscle tone, extremities, and posture. In scoring, each subgroup is evaluated between 0-2 points.
  A minimum of 0 points and a maximum of 16 points are taken from the scale. As the score increases, the baby's stress level increases. Cronbach's alpha coefficient has been reported to be between 0.65-0.81

CONTACTS AND LOCATIONS:
Overall Officials: Emine Serap Çağan, Dr., Study Chair — Ağrı Ibrahim Çeçen University; Eda Akbaş, Midwife, Principal Investigator — Tarsus public hospital; tuğçe sönmez, Dr., Study Chair — Tarsus University
Locations (1):
- Tarsus University, Toroslar, Mersin, Turkey (Türkiye)